CLINICAL TRIAL: NCT04677374
Title: Uptake of Voluntary Medical Male Circumcision Among Men Attending a Sexually Transmitted Infections Clinic in Lilongwe, Malawi
Brief Title: Uptake of Medical Male Circumcision Among Men With Sexually Transmitted Infections
Acronym: VMMC-RITe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-2559; D43TW010060 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-07

CONDITIONS: HIV Infections; Sexually Transmitted Infections
Keywords: Voluntary medical male circumcision; Men with sexually transmitted infections; Uptake; Acceptability; Feasibility
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The intervention will be rolled-out in the implementation phase in a sequential and incremental manner called implementation blocks. Implementation blocks will be as follows: block 1: Intensified health education (I); block 2: Intensified health education and SMS/telephonic Tracing (IT) and finally, Block 3: Intensified health education, SMS/telephonic tracing and transport Reimbursement (RITe)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of care (Placebo Comparator): Participants in this arm will be offered Standard of Care (SOC) referral process for voluntary medical male circumcision (VMMC) services
  Interventions: Other: Standard of care
- Block 1 (intensified health education) (Experimental): Participants in this arm will be offered intensified health education
  Interventions: Behavioral: Intensified Health Education
- Block 2 (intensified health education and SMS/telephonic tracing) (Experimental): Participants in this arm will be offered intensified health education and SMS/telephonic tracing
  Interventions: Behavioral: SMS/telephonic Tracing
- Block 3 (intensified health education, SMS/telephonic tracing and transport reimbursement) (Experimental): Participants in this arm will be offered intensified health education, SMS/telephonic tracing and transport reimbursement
  Interventions: Behavioral: Transportation Reimbursement

INTERVENTIONS:
Other: Standard of care — Standard of care referral approach which is a brief health talk conducted once every morning by a VMMC mobilizer.
  Arms: Standard of care
Behavioral: Intensified Health Education — More detailed health talk conducted during each group health talk session by the VMMC mobilizer and champions describing VMMC, its benefits and how to access the service and testimonies from men who have successfully undergone VMMC
  Arms: Block 1 (intensified health education)
Behavioral: SMS/telephonic Tracing — SMS tracing to remind participants of VMMC appointments
  Arms: Block 2 (intensified health education and SMS/telephonic tracing)
Behavioral: Transportation Reimbursement — Transportation reimbursement to offset the cost of transportation for VMMC appointments
  Arms: Block 3 (intensified health education, SMS/telephonic tracing and transport reimbursement)

SUMMARY:
The intervention includes provision of transport reimbursement for men who will undergo voluntary medical male circumcision (VMMC), intensified health education by a VMMC mobilizer and a male and female VMMC champion and use of a cell phone short messaging service (SMS) and/or telephonic tracing to remind clients of their VMMC appointment (the RITe intervention). The investigators will assess the uptake of VMMC, and acceptability, appropriateness and feasibility of the RITe intervention among uncircumcised men attending a Sexually Transmitted Infection (STI) clinic and health care workers.

This intervention was initially designed to include escorting men interested in circumcision from the STI clinic to a VMMC clinic co-located in the same facility. However, the VMMC clinic space was repurposed to a COVID-19 isolation unit therefore clinic escorts were excluded. In Lieu of clinic escorts, participants will be linked to the nearest health facility of choice where VMMC services are provided by the VMMC mobilizer.

The purpose of the study is to evaluate the impact of using transport reimbursement, intensified health education and SMS/telephonic tracing in increasing the uptake of voluntary medical male circumcision at this clinic.

DETAILED DESCRIPTION:
This study will be a pragmatic, pre- and post-interventional quasi-experimental study combined with a prospective observational study design. The study will have pre-implementation and implementation phases and use a concurrent exploratory mixed method approach.

The study will evaluate the effect of multi-faceted intervention on the uptake of VMMC. The intervention includes use of transport reimbursement for men who will undergo VMMC, Intensified health education by VMMC champions and women and use of SMS/telephonic Tracing to remind clients of their VMMC appointment (the RITe intervention).

The intervention will be conducted in a sequential and incremental manner called implementation blocks. After collecting data from the standard of care period, the first implementation block will be for intensified health education. The next block will combine intensified health education with SMS/telephonic tracing. The last block will combine intensified health education with SMS/telephonic tracing and transport reimbursements. This approach will allow the investigator to compare the effectiveness of different combinations of the strategies in the intervention without necessarily randomizing participants. The sample size for each block is expected to be at least 80 uncircumcised men with STIs. The investigators anticipate that each block may last about 4-12 weeks (to allow the interventions to mature) with one week of no intervention between interventions as a wash out period. However, sample size may be higher if more uncircumcised men present within the minimum 4-week intervention period.

The study population will be men attending the Bwaila STI clinic in Lilongwe Malawi. The study will enroll a minimum of 320 men to depict an uptake rate of circumcision of about 28% (national average including traditional circumcision) among uncircumcised men. However, for each intervention to settle, the investigator will implement each intervention for at least 4 weeks.

Data on uptake of VMMC will be collected through a standardize data collection form in conjunction with routine data from the STI clinic electronic medical registry. Data on acceptability, appropriateness and feasibility will be collected through surveys, interviews and focus group discussions. The investigators will conduct about 280 surveys for acceptability, appropriateness and feasibility with men selected randomly through the implementation period (70 men per intervention block). About 20 in-depth interviews with healthcare workers equally divided by intervention block will be conducted to assess acceptability, appropriateness and feasibility. Finally, the investigators will conduct four focus group discussions with men through the study period to assess acceptability, appropriateness and feasibility of the RITe strategy.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years or older
* Seeking STI care at the Bwaila STI clinic
* Not circumcised
* Healthcare workers at Bwaila STI and VMMC clinic

Exclusion Criteria:

* < 18 years of age

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2242 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Matoga, MD, MSc, Principal Investigator — UNC
Locations (1):
- UNC Project-Malawi (Bwaila District Hospital), Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matoga MM, Kudowa E, Chikuni J, Tsidya M, Tseka J, Ndalama B, Bonongwe N, Mathiya E, Jere E, Yatina D, Kamtambe B, Kapito M, Hosseinipour MC, Chasela CS, Jewett S. Acceptability, feasibility and appropriateness of intensified health education, SMS/phone tracing and transport reimbursement for uptake of voluntary medical male circumcision in a sexually transmitted infections clinic in Malawi: a mixed methods study. medRxiv [Preprint]. 2024 Apr 4:2024.03.27.24304985. doi: 10.1101/2024.03.27.24304985. PMID 38633812
- [Derived] Matoga MM, Kudowa E, Ndalama B, Bonongwe N, Mathiya E, Jere E, Kamtambe B, Chagomerana M, Chasela C, Jewett S, Hosseinipour MC. Effectiveness of an intervention to increase uptake of voluntary medical male circumcision among men with sexually transmitted infections in Malawi: a preinterventional and postinterventional study. BMJ Open. 2023 Oct 3;13(10):e072855. doi: 10.1136/bmjopen-2023-072855. PMID 37788927
- [Derived] Matoga MM, Hosseinipour MC, Jewett S, Chasela C. Uptake of voluntary medical male circumcision among men with sexually transmitted infections in Lilongwe, Malawi: a protocol for a pre-interventional and post-interventional study. BMJ Open. 2022 Jan 18;12(1):e057507. doi: 10.1136/bmjopen-2021-057507. PMID 35042709

RESULTS

PARTICIPANT FLOW:
Groups:
- Block 2 (Intensified Health Education and SMS/Telephonic Tracing): Participants in this arm will be offered intensified health education and short messaging service (SMS)/telephonic tracing
  SMS/telephonic Tracing: SMS tracing to remind participants of VMMC appointments
- Healthcare Workers: Healthcare workers employed at the Sexually Transmitted Infection (STI) clinic who participated in the study
Period: Overall Study
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement) | Healthcare Workers
Started (Healthcare Workers at the participating site who could participate in one or both of the interviews and/or surveys.) | 514 | 731 | 508 | 477 | 12
Completed | 514 | 731 | 508 | 477 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement) | Healthcare Workers | Total
Number analyzed (Participants) | 514 | 731 | 508 | 477 | 12 | 2242
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data reported separately for Male clients and Healthcare Workers.
  years
    Male clients: number analyzed (Participants) | 514 | 731 | 508 | 477 | 0 | 2230
    Male clients | 31 (9) | 30 (8) | 31 (8) | 30 (7) |  | 30 (9)
    Healthcare Workers: number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 12
    Healthcare Workers |  |  |  |  | 37 (7) | 37 (7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not collected for Healthcare Workers.
  Participants
    number analyzed (Participants) | 514 | 731 | 508 | 477 | 0 | 2230
    Female | 0 | 0 | 0 | 0 |  | 0
    Male | 514 | 731 | 508 | 477 |  | 2230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 514 | 731 | 508 | 477 | 12 | 2242
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 514 | 731 | 508 | 477 | 12 | 2242
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 514 | 731 | 508 | 477 | 12 | 2242
Healthcare Workers Years of Experience [Mean (Standard Deviation); unit: Years] — Population: Data not collected for Male clients.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 12 | 12
    (all) |  |  |  |  | 10 (6) | 10 (6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Male Clients Who Will Undergo Circumcision (Uptake of VMMC)
Description: Each participant will be followed for 30 days to determine whether or not they receive circumcision. Number of participants who will undergo circumcision will be reported. The investigators will collect data on the number of participants offered VMMC and the number of participants who will undergo VMMC for each intervention block.
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement)
Number analyzed (Participants) | 514 | 731 | 508 | 477
Participants | 8 | 25 | 13 | 17
Statistical Analysis 1: Comparison: Standard of Care vs Block 1 (Intensified Health Education); Test type: Other; p = 0.044, Test of proportions
Statistical Analysis 2: Comparison: Standard of Care vs Block 2 (Intensified Health Education and SMS/Telephonic Tracing); Test type: Other; p = 0.259, Test of proportions
Statistical Analysis 3: Comparison: Standard of Care vs Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement); Test type: Other; p = 0.044, Test of proportions

2. Primary Outcome: Median Number of Days Taken for Male Clients to Undergo Circumcision From the Day Offered Circumcision at the STI Clinic (Time-to-circumcision)
Description: The duration in days from when participants are offered VMMC to when the participants will undergo VMMC. The investigators will collect data on the number of days taken from the day circumcision is offered for each participant to undergo VMMC through the 30-day Follow-Up period.
Time Frame: up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement)
Number analyzed (Participants) | 8 | 25 | 13 | 17
days | 15 [9 to 18] | 6 [1 to 9] | 3 [0 to 6] | 9 [0 to 14]
Statistical Analysis 1: Comparison: Standard of Care vs Block 1 (Intensified Health Education); Test type: Other; Hazard Ratio (HR) = 2.23, 95% CI 2-sided [1.01 to 4.93]
Statistical Analysis 2: Comparison: Standard of Care vs Block 2 (Intensified Health Education and SMS/Telephonic Tracing); Test type: Other; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [0.69 to 4.00]
Statistical Analysis 3: Comparison: Standard of Care vs Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement); Test type: Other; Hazard Ratio (HR) = 2.31, 95% CI 2-sided [1.00 to 5.36]

3. Secondary Outcome: Percentage of Male Clients Who Reported the RITe Intervention As Acceptable
Description: Acceptability measured quantitatively using the Acceptability of Intervention Measure (AIM) Likert scale surveys. The AIM Likert scale measures acceptability based on four constructs that assess whether an intervention is appealing, likable, welcome and approvable. The AIM score ranges from 6 - 80 1=completely disagree, 2=disagree, 3=Neutral, 4=agree and 5=completely agree. Higher scores indicate agreement with more acceptability items. The percentage is reported for those who strongly agree or agree assessed at Baseline and Follow-Up.
Time Frame: Baseline and Follow-Up, up to 30 days
Population: Participants who received Standard of Care did not participate in the survey. Survey participation was optional for participants in Blocks 1, 2, and 3 and data are reported for all of those who elected to participate. Follow-Up data are missing for some participants who were unavailable.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement)
Number analyzed (Participants) | 0 | 69 | 43 | 34
percentage of participants
  Approve-Baseline |  | 97 | 100 | 100
  Approve-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Approve-Follow-Up |  | 100 | 100 | 100
  Like-Baseline |  | 98.5 | 100 | 97
  Like-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Like-Follow-Up |  | 100 | 97.7 | 96.7
  Welcome-Baseline |  | 97 | 100 | 100
  Welcome-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Welcome-Follow-Up |  | 100 | 97.7 | 100
  Appealing-Baseline |  | 99 | 100 | 97
  Appealing-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Appealing-Follow-Up |  | 100 | 98 | 97

4. Secondary Outcome: Number of Male Clients With Perception That the RITe Intervention is Acceptable
Description: Qualitative assessments for acceptability conducted using focus group discussions with uncircumcised men. Focus group discussions were conducted at Baseline and End of Study Follow Up to complement quantitative findings. Focus group discussions analyzed using thematic analysis and a summary of common themes presented.
Time Frame: Baseline, End of Study Follow Up (approximately Week 82)
Population: Baseline focus group discussions were only conducted in the Standard of Care arm and End of Study Follow Up focus group discussions were conducted only in the Block 3 arm. Focus group discussion participation was limited in number to allow for discussion moderation. Data are reported for all participants who engaged in the discussions.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement)
Number analyzed (Participants) | 16 | 0 | 0 | 11
Participants
  Expressed Liking Intervention-Baseline: number analyzed (Participants) | 16 | 0 | 0 | 0
  Expressed Liking Intervention-Baseline | 14 |  |  |
  Expressed Liking Intervention-End of Study Follow Up: number analyzed (Participants) | 0 | 0 | 0 | 11
  Expressed Liking Intervention-End of Study Follow Up | 0 |  |  | 9
  Expressed Intervention Approval-Baseline: number analyzed (Participants) | 16 | 0 | 0 | 0
  Expressed Intervention Approval-Baseline | 13 |  |  |
  Expressed Intervention Approval-End of Study Follow Up: number analyzed (Participants) | 0 | 0 | 0 | 11
  Expressed Intervention Approval-End of Study Follow Up |  |  |  | 11

5. Secondary Outcome: Percentage of Healthcare Workers Who Rated the RITe Intervention as Feasible
Description: Feasibility measured quantitatively using the Feasibility of Intervention Measure (FIM) Likert scale surveys. The FIM measures feasibility based on four constructs that assess whether an intervention is implementable, possible, resources, and difficult to use. Feasibility assessed among Healthcare Workers only as implementers of the intervention. Surveys for feasibility will be conducted for each intervention block during the implementation phase only. The FIM score range is 5 - 60 with 1=completely disagree, 2=disagree, 3=Neutral, 4=agree and 5=completely agree. Higher scores indicate agreement with more feasibility items. The percentage is reported for those who strongly agree or agree assessed at End of Study Follow Up.
Time Frame: End of Study Follow Up (approximately Week 82)
Population: Data are reported only for Healthcare Workers as this outcome does not apply to Male clients. The Standard of Care arm was not assessed since this outcome focused on the study intervention. Of the 12 participating Healthcare Workers, only 7 were available at the End of Study Follow Up to rate each intervention.
Measure: Number; unit: percentage of Healthcare Workers
Groups:
- Healthcare Workers Standard of Care: Healthcare Workers employed at STI clinic who oversee practices associated with standard of care
- Healthcare Workers Block 1 (Intensified Health Education); Healthcare Workers Block 2 (Intensified Health Education and SMS/Telephonic Tracing): Healthcare Workers employed at STI clinic who implemented intervention
- Healthcare Workers Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement): Healthcare Workers employed at STI clinic who implemented the intervention and participated in the survey
Arm/Group | Healthcare Workers Standard of Care | Healthcare Workers Block 1 (Intensified Health Education) | Healthcare Workers Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Healthcare Workers Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement)
Number analyzed (Participants) | 0 | 7 | 7 | 7
percentage of Healthcare Workers
  Difficult to use |  | 0 | 0 | 0
  Implementable |  | 100 | 100 | 60
  Possible |  | 90 | 100 | 60
  Resources |  | 90 | 0 | 40

6. Secondary Outcome: Number of Healthcare Workers With Perception That the RITe Intervention is Feasible
Description: Qualitative assessments for intervention feasibility conducted using in-depth interviews with Healthcare Workers only at End of Study Follow Up to complement quantitative findings. The interviews were analyzed using thematic analysis and a summary of common themes presented.
Time Frame: End of Study Follow Up (approximately Week 82)
Population: Data are reported only for Healthcare Workers as this outcome does not apply to Male clients. Of the 12 participating Healthcare Workers, only 7 were available for the in-depth interviews at End of Study Follow Up.
Measure: Count of Participants; unit: Participants
Groups:
- Healthcare Workers Standard of Care: Healthcare Workers employed at STI clinic who implemented Standard of Care
- Healthcare Workers Block 1 (Intensified Health Education); Healthcare Workers Block 2 (Intensified Health Education and SMS/Telephonic Tracing): Healthcare Workers employed at STI clinic who implemented the intervention
- Healthcare Workers Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement): Healthcare Workers employed at STI clinic who implemented the intervention and participated in the interviews
Arm/Group | Healthcare Workers Standard of Care | Healthcare Workers Block 1 (Intensified Health Education) | Healthcare Workers Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Healthcare Workers Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement)
Number analyzed (Participants) | 0 | 0 | 0 | 7
Participants
  Concluded Intervention Successfully Implemented |  |  |  | 7
  Concluded Intervention is 'Do-able' |  |  |  | 6

7. Secondary Outcome: Number of Healthcare Workers With Perception That the RITe Intervention is Acceptable at Baseline
Description: Qualitative assessments for acceptability conducted using in-depth interviews with Healthcare Workers at Baseline for the Standard of Care arm to complement quantitative findings. In-depth interviews were analyzed using thematic analysis and a summary of common themes presented.
Time Frame: Baseline
Population: In-depth interview participation was limited in number to allow for discussion moderation. Data are reported for all Healthcare Workers who engaged in the discussions. Of the 12 participating Healthcare Workers, only 10 were available for the in-depth interviews at Baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Healthcare Worker Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement): Healthcare Workers employed at STI clinic who implemented the intervention and participated in interviews
Arm/Group | Healthcare Workers Standard of Care | Healthcare Workers Block 1 (Intensified Health Education) | Healthcare Workers Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Healthcare Worker Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement)
Number analyzed (Participants) | 10 | 0 | 0 | 0
Participants
  Expressed Liking Intervention-Baseline | 9 |  |  |
  Expressed Intervention Approval-Baseline | 10 |  |  |

8. Secondary Outcome: Number of Healthcare Workers With Perception That the RITe Intervention is Acceptable at End of Study Follow Up
Description: Qualitative assessments for acceptability conducted using in-depth interviews with Healthcare Workers at End of Study Follow Up for the Block 3 arm to complement quantitative findings. In-depth interviews were analyzed using thematic analysis and a summary of common themes presented.
Time Frame: End of Study Follow Up (approximately Week 82)
Population: In-depth interview participation was limited in number to allow for discussion moderation. Data are reported for all healthcare workers who engaged in the discussions. Of the 12 participating Healthcare workers, only 7 were available at End of Study Follow Up.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Workers Standard of Care | Healthcare Workers Block 1 (Intensified Health Education) | Healthcare Workers Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Healthcare Worker Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement)
Number analyzed (Participants) | 0 | 0 | 0 | 7
Participants
  Expressed Liking Intervention-End of Study Follow Up |  |  |  | 7
  Expressed Intervention Approval-End of Study Follow Up |  |  |  | 7

9. Secondary Outcome: Percentage of Male Clients Who Reported the RITe Intervention As Appropriate
Description: Appropriateness measured quantitatively using the Intervention Appropriateness Measure (IAM) Likert scale surveys. The IAM Likert scale measures appropriateness based on four constructs that assess whether an intervention is embarrassing, culturally & religiously suitable, and a good idea. Surveys for appropriateness were conducted at baseline and during implementation of each intervention block. The IAM score range is 5 - 85 from a scale with 1=completely disagree, 2=disagree, 3=Neutral, 4=agree and 5=completely agree. Higher scores indicate agreement with more appropriateness items. The percentage is reported for those who strongly agree or agree assessed at Baseline and Follow-Up.
Time Frame: Baseline and Follow-Up, up to 30 days
Population: Participants who received Standard of Care did not participate in the survey. Survey participation was optional and data are reported for all of those who elected to participate. Follow-Up data are missing for some participants who were unavailable.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement)
Number analyzed (Participants) | 0 | 69 | 43 | 34
percentage of participants
  Culturally suitable-Baseline |  | 62.3 | 27.9 | 11.8
  Culturally suitable-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Culturally suitable-Follow-Up |  | 42.1 | 100 | 100
  Embarrassing-Baseline |  | 26.1 | 9.3 | 2.9
  Embarrassing-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Embarrassing-Follow-Up |  | 31.6 | 0 | 0
  Good idea-Baseline |  | 98.6 | 100 | 100
  Good idea-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Good idea-Follow-Up |  | 100 | 100 | 100
  Religiously suitable-Baseline |  | 63.8 | 98 | 11.8
  Religiously suitable-Follow-Up: number analyzed (Participants) | 0 | 59 | 43 | 30
  Religiously suitable-Follow-Up |  | 42.1 | 93 | 96.7

10. Secondary Outcome: Number of Male Clients With Perception That the RITe Intervention is Appropriate
Description: Qualitative assessments for appropriateness conducted using focus group discussions with uncircumcised men. Focus group discussions conducted at Baseline and End of Study Follow Up to complement quantitative findings. Focus group discussions were analyzed using thematic analysis and a summary of common themes presented.
Time Frame: Baseline, End of Study Follow Up (approximately Week 82)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement)
Number analyzed (Participants) | 16 | 0 | 0 | 11
Participants
  Expressed that Intervention is a Good Idea-Baseline: number analyzed (Participants) | 16 | 0 | 0 | 0
  Expressed that Intervention is a Good Idea-Baseline | 15 |  |  |
  Expressed that Intervention is a Good Idea-End of Study Follow Up: number analyzed (Participants) | 0 | 0 | 0 | 11
  Expressed that Intervention is a Good Idea-End of Study Follow Up |  |  |  | 11
  Intervention Aligned with Religion-Baseline: number analyzed (Participants) | 16 | 0 | 0 | 0
  Intervention Aligned with Religion-Baseline | 13 |  |  |
  Intervention Aligned with Religion-End of Study Follow Up: number analyzed (Participants) | 0 | 0 | 0 | 11
  Intervention Aligned with Religion-End of Study Follow Up |  |  |  | 10
  Intervention Aligned with Culture-Baseline: number analyzed (Participants) | 16 | 0 | 0 | 0
  Intervention Aligned with Culture-Baseline | 11 |  |  |
  Intervention Aligned with Culture-End of Study Follow Up: number analyzed (Participants) | 0 | 0 | 0 | 11
  Intervention Aligned with Culture-End of Study Follow Up |  |  |  | 11

11. Secondary Outcome: Number of Healthcare Workers With Perception That the RITe Intervention is Appropriate at Baseline
Description: Qualitative assessments for appropriateness conducted using in-depth interviews with Healthcare Workers only. The interviews were conducted at Baseline to complement quantitative findings. The Interviews were analyzed using thematic analysis and a summary of common themes presented.
Time Frame: Baseline
Population: Baseline in-depth interviews were only conducted in the Standard of Care arm. In-depth interview participation was limited to Healthcare Workers who accepted to participate and who engaged in the discussions. Of the 12 participating Healthcare Workers, only 10 were available at Baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Healthcare Worker Standard of Care: Healthcare Workers employed at STI clinic who oversee practices associated with standard of care
- Healthcare Worker Block 1 (Intensified Health Education); Healthcare Worker Block 2 (Intensified Health Education and SMS/Telephonic Tracing): Healthcare Workers employed at STI clinic who implemented the intervention
- Healthcare Worker Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement): Healthcare Workers employed at STI clinic who implemented the intervention and participated in the interviews
Arm/Group | Healthcare Worker Standard of Care | Healthcare Worker Block 1 (Intensified Health Education) | Healthcare Worker Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Healthcare Worker Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement)
Number analyzed (Participants) | 10 | 0 | 0 | 0
Participants
  Expressed that Intervention is a Good Idea-Baseline | 10 |  |  |
  Intervention Aligned with Religion-Baseline | 8 |  |  |
  Intervention Aligned with Culture-Baseline | 8 |  |  |

12. Secondary Outcome: Number of Healthcare Workers With Perception That the RITe Intervention is Appropriate at End of Study Follow Up
Description: Qualitative assessments for appropriateness conducted using in-depth interviews with Healthcare Workers only. The interviews were conducted at End of Study Follow Up to complement quantitative findings. The Interviews were analyzed using thematic analysis and a summary of common themes presented.
Time Frame: End of Study Follow Up (approximately Week 82)
Population: These in-depth interviews were conducted only in the Block 3 arm with participation limited to Healthcare Workers who accepted to participate. Data are reported for those who engaged in the discussions. Of the 12 participating Healthcare Workers, only 7 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthcare Worker Standard of Care | Healthcare Worker Block 1 (Intensified Health Education) | Healthcare Worker Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Healthcare Worker Block 3 (Intensified Health Education, SMS/Tracing and Transport Reimbursement)
Number analyzed (Participants) | 0 | 0 | 0 | 7
Participants
  Expressed that Intervention is a Good Idea-End of Study Follow Up |  |  |  | 7
  Intervention Aligned with Religion-End of Study Follow Up |  |  |  | 7
  Intervention Aligned with Culture-End of Study Follow Up |  |  |  | 7

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent at Week 0 up to 30 days afterwards.
Description: Adverse events were not collected for Healthcare Workers.
Arm/Group | Standard of Care | Block 1 (Intensified Health Education) | Block 2 (Intensified Health Education and SMS/Telephonic Tracing) | Block 3 (Intensified Health Education, SMS/Telephonic Tracing and Transport Reimbursement)
All-Cause Mortality (participants affected / at risk) | 0/514 | 0/731 | 0/508 | 0/477
Serious Adverse Events (participants affected / at risk) | 0/514 | 0/731 | 0/508 | 0/477
Other Adverse Events (participants affected / at risk) | 0/514 | 0/731 | 0/508 | 0/477

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT04677374/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT04677374/ICF_001.pdf